CLINICAL TRIAL: NCT01037881
Title: A Phase 2, Proof of Concept and Dose Finding Study, Investigating Treatment Efficacy of LEO 29102 Cream, LEO 29102 Cream Vehicle, and Elidel® Cream 10 mg/g, After Cutaneous Administration Twice Daily for 4 Weeks
Brief Title: LEO 29102 Cream in the Treatment of Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LEO 29102-C21; EudraCT Number 2009-013792-22 (Registry Identifier: European Clinical Trials Database)
Record Dates: First submitted 2009-12-21; First posted 2009-12-23 (Estimated); Results first posted 2019-10-14 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2018-08

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — 2-(6-(2-(3,5-dichloro-4-pyridyl)acetyl)-2,3-dimethoxyphenoxy)-N-propylacetamide; pimecrolimus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- LEO 29102 0.03 mg/g cream (Experimental)
  Interventions: Drug: LEO 29102
- LEO 29102 0.1 mg/g cream (Experimental)
  Interventions: Drug: LEO 29102
- LEO 29102 0.3 mg/g cream (Experimental)
  Interventions: Drug: LEO 29102
- LEO 29102 1.0 mg/g cream (Experimental)
  Interventions: Drug: LEO 29102
- LEO 29102 2.5 mg/g cream (Experimental)
  Interventions: Drug: LEO 29102
- LEO 29102 cream vehicle (Placebo Comparator)
  Interventions: Drug: LEO 29102
- Elidel® cream (pimecrolimus) 10 mg/g (Active Comparator)
  Interventions: Drug: Elidel®

INTERVENTIONS:
Drug: LEO 29102 — comparison of different dosages of drug
  Arms: LEO 29102 0.03 mg/g cream; LEO 29102 0.1 mg/g cream; LEO 29102 0.3 mg/g cream; LEO 29102 1.0 mg/g cream; LEO 29102 2.5 mg/g cream; LEO 29102 cream vehicle
Drug: Elidel® — comparison
  Arms: Elidel® cream (pimecrolimus) 10 mg/g

SUMMARY:
This is a proof of concept and dose finding Phase II trial comparing 5 dose strengths with vehicle and an active comparator (Elidel cream 10 mg/g) in a 4 week, twice daily treatment regimen in mild to moderate atopic dermatitis patients.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of atopic dermatitis defined according to Hanifin and Rajka
* IGA assessment scored as mild (2) to moderate (3) atopic dermatitis
* Treatment lesions located on the trunk and limbs
* Treatment lesions involving 3% to 10% of the total body surface area
* Patients of either gender between 18 years and 65 years of age

Exclusion Criteria:

* Systemic treatment with immunosuppressive drugs or corticosteroids within 6 weeks prior to randomisation
* Topical treatment with immunomodulators (pimecrolimus, tacrolimus) within 2 weeks prior to randomisation
* Topical treatment with corticosteroids from WHO groups II, III or IV within 1 week prior to randomisation
* Use of topical or systemic antibiotics within 2 weeks prior to randomisation
* PUVA or UVB therapy within 4 weeks prior to randomisation
* Clinical infection (viral, fungal or bacterial) on the treatment area
* Known or suspected severe renal insufficiency or severe hepatic disorders
* Patients with history of an immunocompromised disease (e.g., lymphoma, HIV, Wiskott-Aldrich Syndrome)
* Patients with concomitant serious disease (e.g., cancer) which might affect the AD treatment in this trial
* Females who are pregnant or are breast feeding
* Females intending to temporarily or permanently stop their hormonal contraceptive regime during and up to one month post study termination visit

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2009-12; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Expert, Study Director — LEO Pharma
Locations (3):
- Windsor Clinical Research Inc., Windsor, Ontario, Canada
- Helsinki University Central Hospital, Helsinki, Finland
- Klinik und Poliklinik für Dermatologie, Universität Bonn, Bonn, Germany

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants received investigational medicinal products for up to 4-weeks followed by a 28 day follow-up period.
Groups:
- LEO 29102 Vehicle: LEO 29102 cream vehicle applied topically twice daily - in the morning and in the evening - on a total area of 3-10% of the total body surface area (BSA) for up to 4 weeks. Participants who were evaluated by the investigator to be symptom-free (as defined by an investigator's global assessment [IGA] of 0 or 1, i.e. clear or almost clear of symptoms) at any of Visits 2(Day 7), 3(Day 14) or 4(Day 21) could stop treatment at the investigator's discretion. They were to remain in the study and attend all visits up to and including Visit 6 (Day 56). The participants had to have study medication dispensed and should restart treatment if required, based on the participant's own judgement. More than one discontinuation/restart cycle was allowed.
- LEO 29102 0.03 mg/g: LEO 29102 0.03 mg/g cream applied topically twice daily - in the morning and in the evening - on a total area of 3-10% of the total BSA for up to 4 weeks. Participants who were evaluated by the investigator to be symptom-free (as defined by an IGA of 0 or 1, i.e. clear or almost clear of symptoms) at any of Visits 2(Day 7), 3(Day 14) or 4(Day 21) could stop treatment at the investigator's discretion. They were to remain in the study and attend all visits up to and including Day 56. The participants had to have study medication dispensed and should restart treatment if required, based on the participant's own judgement. More than one discontinuation/restart cycle was allowed.
- LEO 29102 0.1 mg/g: LEO 29102 0.1 mg/g cream applied topically twice daily - in the morning and in the evening - on a total area of 3-10% of the total BSA for up to 4 weeks. Participants who were evaluated by the investigator to be symptom-free (as defined by an IGA of 0 or 1) at any of Visits 2(Day 7), 3(Day 14) or 4(Day 21) could stop treatment at the investigator's discretion. They were to remain in the study and attend all visits up to and including Day 56. The participants had to have study medication dispensed and should restart treatment if required, based on the participant's own judgement. More than one discontinuation/restart cycle was allowed.
- LEO 29102 0.3 mg/g: LEO 29102 0.3 mg/g cream applied topically twice daily - in the morning and in the evening - on a total area of 3-10% of the total BSA for up to 4 weeks. Participants who were evaluated by the investigator to be symptom-free (as defined by an IGA of 0 or 1) at any of Visits 2(Day 7), 3(Day 14) or 4(Day 21) could stop treatment at the investigator's discretion. They were to remain in the study and attend all visits up to and including Day 56. The participants had to have study medication dispensed and should restart treatment if required, based on the participant's own judgement. More than one discontinuation/restart cycle was allowed.
- LEO 29102 1.0 mg/g: LEO 29102 1.0 mg/g cream applied topically twice daily - in the morning and in the evening - on a total area of 3-10% of the total BSA for up to 4 weeks. Participants who were evaluated by the investigator to be symptom-free (as defined by an IGA of 0 or 1) at any of Visits 2(Day 7), 3(Day 14) or 4(Day 21) could stop treatment at the investigator's discretion. They were to remain in the study and attend all visits up to and including Day 56. The participant had to have study medication dispensed and should restart treatment if required, based on the participant's own judgement. More than one discontinuation/restart cycle was allowed.
  Participants were not randomized to this treatment until the results from the hormone screen blood samples from at least 10 participants in each of the five initial treatment arms (LEO 29102 0.03 mg/g cream, 0.1 mg/g cream,0.3 mg/g cream, cream vehicle, and Elidel®) were available and no safety concerns had been raised.
- LEO 29102 2.5 mg/g: LEO 29102 2.5 mg/g cream applied topically twice daily - in the morning and in the evening - on a total area of 3-10% of the total BSA for up to 4 weeks. Participants who were evaluated by the investigator to be symptom-free (as defined by an IGA of 0 or 1) at any of Visits 2(Day 7), 3(Day 14) or 4(Day 21) could stop treatment at the investigator's discretion. They were to remain in the study and attend all visits up to and including Day 56. The participants had to have study medication dispensed and should restart treatment if required, based on the participant's own judgement. More than one discontinuation/restart cycle was allowed.
  Participants were not randomized to this treatment until the results from the hormone screen blood samples from at least 10 participants in each of the five initial treatment arms (LEO 29102 0.03 mg/g cream, 0.1 mg/g cream,0.3 mg/g cream, cream vehicle, and Elidel®) were available and no safety concerns had been raised.
- Elidel® 10 mg/g: Elidel® applied topically twice daily - in the morning and in the evening - on a total area of 3-10% of the total BSA for up to 4 weeks.
  Participants who were evaluated by the investigator to be symptom-free (as defined by an IGA of 0 or 1) at any of Visits 2(Day 7), 3(Day 14) or 4(Day 21) could stop treatment at the investigator's discretion. They were to remain in the study and attend all visits up to and including Day 56. The participants had to have study medication dispensed and should restart treatment if required, based on the participant's own judgement. More than one discontinuation/restart cycle was allowed.
Period: Overall Study
Arm/Group | LEO 29102 Vehicle | LEO 29102 0.03 mg/g | LEO 29102 0.1 mg/g | LEO 29102 0.3 mg/g | LEO 29102 1.0 mg/g | LEO 29102 2.5 mg/g | Elidel® 10 mg/g
Started | 25 | 24 | 25 | 25 | 29 | 30 | 25
Completed | 19 | 22 | 22 | 24 | 26 | 27 | 23
Not Completed | 6 | 2 | 3 | 1 | 3 | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- LEO 29102 Vehicle: Treatment with LEO 29102 cream vehicle twice daily - in the morning and in the evening - for up to 4 weeks
- LEO 29102 0.03 mg/g: Treatment with LEO 29102 0.03 mg/g cream twice daily - in the morning and in the evening - for up to 4 weeks
- LEO 29102 0.1 mg/g: Treatment with LEO 29102 0.1 mg/g cream twice daily - in the morning and in the evening - for up to 4 weeks
- LEO 29102 0.3 mg/g: Treatment with LEO 29102 0.3 mg/g cream twice daily - in the morning and in the evening - for up to 4 weeks
- LEO 29102 1.0 mg/g: Treatment with LEO 29102 1.0 mg/g cream twice daily - in the morning and in the evening - for up to 4 weeks
- LEO 29102 2.5 mg/g: Treatment with LEO 29102 2.5 mg/g cream twice daily - in the morning and in the evening - for up to 4 weeks
- Elidel® 10 mg/g: Treatment with Elidel® twice daily - in the morning and in the evening - for up to 4 weeks
- Total: Total of all reporting groups
Arm/Group | LEO 29102 Vehicle | LEO 29102 0.03 mg/g | LEO 29102 0.1 mg/g | LEO 29102 0.3 mg/g | LEO 29102 1.0 mg/g | LEO 29102 2.5 mg/g | Elidel® 10 mg/g | Total
Number analyzed (Participants) | 25 | 24 | 25 | 25 | 29 | 30 | 25 | 183
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.1 (14.0) | 36.2 (14.4) | 34.9 (11.8) | 38.3 (12.6) | 32.0 (10.0) | 35.5 (13.7) | 29.9 (8.8) | 35.1 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 8 | 10 | 4 | 15 | 13 | 9 | 70
  Male | 14 | 16 | 15 | 21 | 14 | 17 | 16 | 113
Region of Enrollment [Number; unit: participants]
  Canada | 4 | 6 | 5 | 6 | 6 | 6 | 4 | 37
  Finland | 3 | 0 | 2 | 2 | 6 | 6 | 3 | 22
  Germany | 18 | 18 | 18 | 17 | 17 | 18 | 18 | 124

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change in Eczema Area and Severity Index (EASI) Score From Baseline (Last Observation Carried Forward [LOCF])
Description: The EASI is a composite score based on the evaluation of four characteristic atopic dermatitis (AD) signs and symptoms; erythema, oedema/induration/papulation, excoriation and lichenification together with the area involved.
  For each body region, the investigator rated four clinical signs of AD using the following severity scale:
  0 = none/absent
  1. = mild
  2. = moderate
  3. = severe
  The EASI score ranges from 0-12, a higher score equals a worse outcome. Baseline was defined as Day 0. Mean values in table are least squares mean adjusted for the effect of (pooled) country.
Time Frame: Baseline (Day 0) and end of treatment (Day 28)
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Groups:
- LEO 29102 2.5 mg/g: Treatment with LEO 29102 2.5 mg/g cream twice daily - in the morning and in the evening - for up to 4 week
Arm/Group | LEO 29102 Vehicle | LEO 29102 0.03 mg/g | LEO 29102 0.1 mg/g | LEO 29102 0.3 mg/g | LEO 29102 1.0 mg/g | LEO 29102 2.5 mg/g | Elidel® 10 mg/g
Number analyzed (Participants) | 25 | 24 | 25 | 25 | 29 | 30 | 25
units on a scale | -0.85 (6.85) | -2.13 (3.00) | -1.09 (5.81) | -2.86 (2.99) | -2.41 (2.38) | -2.50 (3.28) | -3.30 (2.51)
Statistical Analysis 1: Comparison: LEO 29102 Vehicle vs LEO 29102 0.03 mg/g; Active treatment minus vehicle, adjusted for the effect of (pooled) country; Test type: Superiority; p = 0.27, ANOVA; Difference in least squares mean = -1.29, 95% CI 2-sided [-3.60 to 1.03]
Statistical Analysis 2: Comparison: LEO 29102 Vehicle vs LEO 29102 0.1 mg/g; Active treatment minus vehicle, adjusted for the effect of (pooled) country; Test type: Superiority; p = 0.83, ANOVA; Difference in least squares mean = -0.25, 95% CI 2-sided [-2.53 to 2.04]
Statistical Analysis 3: Comparison: LEO 29102 Vehicle vs LEO 29102 0.3 mg/g; Active treatment minus vehicle, adjusted for the effect of (pooled) country; Test type: Superiority; p = 0.08, ANOVA; Difference in least squares mean = -2.01, 95% CI 2-sided [-4.30 to 0.28]
Statistical Analysis 4: Comparison: LEO 29102 Vehicle vs LEO 29102 1.0 mg/g; Active treatment minus vehicle, adjusted for the effect of (pooled) country; Test type: Superiority; p = 0.16, ANOVA; Difference in least squares mean = -1.56, 95% CI 2-sided [-3.77 to 0.65]
Statistical Analysis 5: Comparison: LEO 29102 Vehicle vs LEO 29102 2.5 mg/g; Active treatment minus vehicle, adjusted for the effect of (pooled) country; Test type: Superiority; p = 0.14, ANOVA; Difference in least squares mean = -1.65, 95% CI 2-sided [-3.84 to 0.54]
Statistical Analysis 6: Comparison: LEO 29102 Vehicle vs Elidel® 10 mg/g; Active treatment minus vehicle, adjusted for the effect of (pooled) country; Test type: Superiority; p = 0.04, ANOVA; Difference in least squares mean = -2.46, 95% CI 2-sided [-4.47 to -0.17]
Statistical Analysis 7: Comparison: LEO 29102 Vehicle vs Elidel® 10 mg/g; LEO 29102 treatment minus Elidel, adjusted for the effect of (pooled) country; Test type: Superiority; p = 0.04, ANOVA; Difference in least squares mean = 2.46, 95% CI 2-sided [0.17 to 4.74]
Statistical Analysis 8: Comparison: LEO 29102 0.03 mg/g vs Elidel® 10 mg/g; LEO 29102 treatment minus Elidel, adjusted for the effect of (pooled) country; Test type: Superiority; p = 0.32, ANOVA; Difference in least squares mean = 1.17, 95% CI 2-sided [-1.14 to 3.48]
Statistical Analysis 9: Comparison: LEO 29102 0.1 mg/g vs Elidel® 10 mg/g; LEO 29102 treatment minus Elidel, adjusted for the effect of (pooled) country; Test type: Superiority; p = 0.06, ANOVA; Difference in least squares mean = 2.21, 95% CI 2-sided [-0.08 to 4.50]
Statistical Analysis 10: Comparison: LEO 29102 0.3 mg/g vs Elidel® 10 mg/g; LEO 29102 treatment minus Elidel, adjusted for the effect of (pooled) country; Test type: Superiority; p = 0.70, ANOVA; Difference in least squares mean = 0.45, 95% CI 2-sided [-1.84 to 2.73]
Statistical Analysis 11: Comparison: LEO 29102 1.0 mg/g vs Elidel® 10 mg/g; LEO 29102 treatment minus Elidel, adjusted for the effect of (pooled) country; Test type: Superiority; p = 0.42, ANOVA; Difference in least squares mean = 0.90, 95% CI 2-sided [-1.31 to 3.10]
Statistical Analysis 12: Comparison: LEO 29102 2.5 mg/g vs Elidel® 10 mg/g; LEO 29102 treatment minus Elidel, adjusted for the effect of (pooled) country; Test type: Superiority; p = 0.47, ANOVA; Difference in least squares mean = 0.81, 95% CI 2-sided [-1.38 to 3.00]

2. Secondary Outcome: Number of Participants That Were Symptom Free Responders (LOCF)
Description: The IGA (Investigator's global assessment) of disease severity on the body (trunk and limbs excluding the hands) was assessed based on visual evaluation by use of the following definitions of severity:
  0. Clear - no inflammatory signs of AD
  1. Almost clear - just perceptible erythema, and just perceptible papulation/infiltration
  2. Mild - mild erythema, and mild papulation/infiltration
  3. Moderate - moderate erythema, and moderate papulation/infiltration
  4. Severe - severe erythema, and-severe papulation/infiltration
  5. Very severe - severe erythema, and severe papulation/infiltration with oozing/crusting.
  Symptom free responders were defined as an IGA of 0 (Clear) or 1 (Almost clear) at the end of treatment.
Time Frame: At end of treatment (Day 28)
Measure: Count of Participants; unit: Participants
Arm/Group | LEO 29102 Vehicle | LEO 29102 0.03 mg/g | LEO 29102 0.1 mg/g | LEO 29102 0.3 mg/g | LEO 29102 1.0 mg/g | LEO 29102 2.5 mg/g | Elidel® 10 mg/g
Number analyzed (Participants) | 25 | 24 | 25 | 25 | 29 | 30 | 25
Participants
  Responder | 6 | 2 | 5 | 9 | 10 | 13 | 12
  Non-responder | 19 | 22 | 20 | 16 | 19 | 17 | 13

3. Secondary Outcome: Participants' Assessment of Pruritus on Trunk and Limbs
Description: Participants' assessment of pruritus on trunk and limbs was assessed at end of treatment by use of the scale below.
  * Absent - no itching
  * Mild - occasional, slight itching
  * Moderate - constant or intermittent itching which is not disturbing sleep
  * Severe - intolerable itching which is disturbing sleep
  The assessment was based on the average degree of pruritus over the last 24 hours.
Time Frame: At end of treatment (Day 28)
Measure: Count of Participants; unit: Participants
Groups:
- Elidel®10 mg/g: Treatment with Elidel® twice daily - in the morning and in the evening - for up to 4 weeks
Arm/Group | LEO 29102 Vehicle | LEO 29102 0.03 mg/g | LEO 29102 0.1 mg/g | LEO 29102 0.3 mg/g | LEO 29102 1.0 mg/g | LEO 29102 2.5 mg/g | Elidel®10 mg/g
Number analyzed (Participants) | 25 | 24 | 25 | 25 | 29 | 30 | 25
Participants
  Absent | 5 | 1 | 4 | 7 | 5 | 7 | 6
  Mild | 8 | 7 | 9 | 7 | 15 | 13 | 14
  Moderate | 8 | 9 | 9 | 11 | 8 | 6 | 4
  Severe | 4 | 7 | 3 | 0 | 1 | 4 | 1

4. Secondary Outcome: Participants' Overall Assessment of Disease Severity
Description: Participants' overall assessment of disease severity on trunk and limbs (excluding the hands) was assessed at end of treatment by use of the following scale: clear, very mild, mild, moderate, severe.
  The assessment was based on the condition of the disease at the time of the evaluation and not in relation to the condition at a previous visit.
Time Frame: At end of treatment (Day 28)
Measure: Count of Participants; unit: Participants
Arm/Group | LEO 29102 Vehicle | LEO 29102 0.03 mg/g | LEO 29102 0.1 mg/g | LEO 29102 0.3 mg/g | LEO 29102 1.0 mg/g | LEO 29102 2.5 mg/g | Elidel® 10 mg/g
Number analyzed (Participants) | 25 | 24 | 25 | 25 | 29 | 30 | 25
Participants
  Clear | 2 | 1 | 2 | 3 | 4 | 1 | 2
  Very mild | 5 | 1 | 4 | 5 | 5 | 12 | 11
  Mild | 8 | 10 | 9 | 5 | 10 | 10 | 8
  Moderate | 6 | 9 | 7 | 11 | 10 | 4 | 3
  Severe | 4 | 3 | 3 | 1 | 0 | 3 | 1

5. Secondary Outcome: Number of Participants That Were Symptom Free Responders by Visit
Description: Symptom free responders were defined as an IGA of 0 (Clear) or 1 (Almost clear) according to Investigator's global assessment of disease severity on trunk and limbs at the end of treatment.
Time Frame: At Visit 2 (Day 7), Visit 3 (Day 14), Visit 4 (Day 21) and end of treatment (Day 28)
Population: Occurrences of early withdrawal, non-compliance, prohibited medication, missing application of study medication and participants missing visits resulted in not all participants being analyzed at all visits.
Measure: Count of Participants; unit: Participants
Arm/Group | LEO 29102 Vehicle | LEO 29102 0.03 mg/g | LEO 29102 0.1 mg/g | LEO 29102 0.3 mg/g | LEO 29102 1.0 mg/g | LEO 29102 2.5 mg/g | Elidel® 10 mg/g
Number analyzed (Participants) | 25 | 24 | 25 | 25 | 29 | 30 | 25
Participants
  Visit 2 (Day 7): number analyzed (Participants) | 25 | 23 | 25 | 24 | 28 | 30 | 25
  Visit 2 (Day 7): Responder | 2 | 1 | 2 | 1 | 5 | 5 | 2
  Visit 2 (Day 7): Non-responder | 23 | 22 | 23 | 23 | 23 | 25 | 23
  Visit 3 (Day 14): number analyzed (Participants) | 21 | 24 | 23 | 24 | 27 | 29 | 24
  Visit 3 (Day 14): Responder | 4 | 1 | 3 | 3 | 5 | 7 | 8
  Visit 3 (Day 14): Non-responder | 17 | 23 | 20 | 21 | 22 | 22 | 16
  Visit 4 (Day 21): number analyzed (Participants) | 20 | 22 | 23 | 23 | 25 | 27 | 23
  Visit 4 (Day 21): Responder | 4 | 2 | 6 | 7 | 5 | 11 | 8
  Visit 4 (Day 21): Non-responder | 16 | 20 | 17 | 16 | 20 | 16 | 15
  Visit 5 (Day 28): number analyzed (Participants) | 19 | 22 | 22 | 24 | 26 | 27 | 23
  Visit 5 (Day 28): Responder | 6 | 2 | 5 | 9 | 10 | 12 | 12
  Visit 5 (Day 28): Non-responder | 13 | 20 | 17 | 15 | 16 | 15 | 11

6. Secondary Outcome: Absolute Change in Eczema Area and Severity Index (EASI) Score From Baseline by Visit
Description: as for outcome 1
Time Frame: Baseline and at Visit 2 (Day 7), Visit 3 (Day 14), Visit 4 (Day 21)
Population: Data was tabulated using an observed cases approach and therefore only contains data from participants who attended the specific visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LEO 29102 Vehicle | LEO 29102 0.03 mg/g | LEO 29102 0.1 mg/g | LEO 29102 0.3 mg/g | LEO 29102 1.0 mg/g | LEO 29102 2.5 mg/g | Elidel® 10 mg/g
Number analyzed (Participants) | 25 | 24 | 25 | 25 | 29 | 30 | 25
units on a scale
  Visit 2 (Day 7): number analyzed (Participants) | 25 | 23 | 25 | 24 | 28 | 30 | 25
  Visit 2 (Day 7) | -0.09 (5.27) | -1.26 (1.72) | -0.93 (1.82) | -1.43 (2.53) | -1.64 (1.71) | -1.48 (2.28) | -1.21 (2.17)
  Visit 3 (Day 14): number analyzed (Participants) | 21 | 24 | 23 | 24 | 27 | 29 | 24
  Visit 3 (Day 14) | -1.77 (2.77) | -1.48 (2.19) | -1.30 (2.28) | -2.19 (3.14) | -1.67 (2.15) | -1.52 (3.17) | -1.82 (2.39)
  Visit 4 (Day 21): number analyzed (Participants) | 20 | 22 | 23 | 23 | 25 | 27 | 23
  Visit 4 (Day 21) | -1.62 (4.18) | -1.76 (2.67) | -0.89 (5.94) | -2.21 (3.27) | -1.90 (2.57) | -2.53 (2.18) | -2.16 (2.22)

ADVERSE EVENTS:
Time Frame: From baseline (Day 0) to Day 28±3 (end of treatment) and follow-up phase (from end of treatment to Day 56±4)
Description: The Safety Analysis Set only consisted of participants who applied study medication. One participant from the LEO 29102 1.0 mg/g arm, did not apply any study medication and was therefore excluded from the safety analysis.
Groups:
- LEO 29102 Cream Vehicle - Treatment Phase; LEO 29102 Cream Vehicle - Follow-up Phase: Treatment with LEO 29102 cream vehicle twice daily - in the morning and in the evening - for up to 4 weeks
- LEO 29102 0.03 mg/g Cream - Treatment Phase; LEO 29102 0.03 mg/g Cream - Follow-up Phase: Treatment with LEO 29102 0.03 mg/g cream twice daily - in the morning and in the evening - for up to 4 weeks
- LEO 29102 0.1 mg/g Cream - Treatment Phase; LEO 29102 0.1 mg/g Cream - Follow-up Phase: Treatment with LEO 29102 0.1 mg/g cream twice daily - in the morning and in the evening - for up to 4 weeks
- LEO 29102 0.3 mg/g Cream - Treatment Phase; LEO 29102 0.3 mg/g Cream - Follow-up Phase: Treatment with LEO 29102 0.3 mg/g cream twice daily - in the morning and in the evening - for up to 4 weeks
- LEO 29102 1.0 mg/g Cream - Treatment Phase; LEO 29102 1.0 mg/g Cream - Follow-up Phase: Treatment with LEO 29102 1.0 mg/g cream twice daily - in the morning and in the evening - for up to 4 weeks
- LEO 29102 2.5 mg/g Cream - Treatment Phase; LEO 29102 2.5 mg/g Cream - Follow-up Phase: Treatment with LEO 29102 2.5 mg/g cream twice daily - in the morning and in the evening - for up to 4 weeks
- Elidel® Cream (Pimecrolimus) 10 mg/g - Treatment Phase; Elidel® 10 mg/g - Follow-up Phase: Treatment with Elidel® twice daily - in the morning and in the evening - for up to 4 weeks
Arm/Group | LEO 29102 Cream Vehicle - Treatment Phase | LEO 29102 0.03 mg/g Cream - Treatment Phase | LEO 29102 0.1 mg/g Cream - Treatment Phase | LEO 29102 0.3 mg/g Cream - Treatment Phase | LEO 29102 1.0 mg/g Cream - Treatment Phase | LEO 29102 2.5 mg/g Cream - Treatment Phase | Elidel® Cream (Pimecrolimus) 10 mg/g - Treatment Phase | LEO 29102 Cream Vehicle - Follow-up Phase | LEO 29102 0.03 mg/g Cream - Follow-up Phase | LEO 29102 0.1 mg/g Cream - Follow-up Phase | LEO 29102 0.3 mg/g Cream - Follow-up Phase | LEO 29102 1.0 mg/g Cream - Follow-up Phase | LEO 29102 2.5 mg/g Cream - Follow-up Phase | Elidel® 10 mg/g - Follow-up Phase
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/24 | 0/25 | 0/25 | 0/28 | 0/30 | 0/25 | 0/25 | 0/24 | 0/25 | 0/25 | 0/28 | 0/30 | 0/25
Other Adverse Events (participants affected / at risk) | 13/25 | 11/24 | 8/25 | 8/25 | 8/28 | 8/30 | 8/25 | 1/25 | 0/24 | 2/25 | 0/25 | 2/28 | 4/30 | 2/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LEO 29102 Cream Vehicle - Treatment Phase (N=25) | LEO 29102 0.03 mg/g Cream - Treatment Phase (N=24) | LEO 29102 0.1 mg/g Cream - Treatment Phase (N=25) | LEO 29102 0.3 mg/g Cream - Treatment Phase (N=25) | LEO 29102 1.0 mg/g Cream - Treatment Phase (N=28) | LEO 29102 2.5 mg/g Cream - Treatment Phase (N=30) | Elidel® Cream (Pimecrolimus) 10 mg/g - Treatment Phase (N=25) | LEO 29102 Cream Vehicle - Follow-up Phase (N=25) | LEO 29102 0.03 mg/g Cream - Follow-up Phase (N=24) | LEO 29102 0.1 mg/g Cream - Follow-up Phase (N=25) | LEO 29102 0.3 mg/g Cream - Follow-up Phase (N=25) | LEO 29102 1.0 mg/g Cream - Follow-up Phase (N=28) | LEO 29102 2.5 mg/g Cream - Follow-up Phase (N=30) | Elidel® 10 mg/g - Follow-up Phase (N=25)
Conjunctivitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis allergic (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Keratitis (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Application site irritation (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Application site pain (General disorders) | 0 | 2 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Application site pruritus (General disorders) | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Application site vesicles (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fungal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Herpes simplex ophthalmic (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 2 | 0 | 2 | 2 | 1 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Burning sensation (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Breast swelling (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholestatic pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 3 | 1 | 3 | 0 | 1 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Knee operation (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Osteotomy (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Local swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Arthroscopy (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Company acknowledges the investigators' right to publish the entire results of the study, irrespective of outcome. The Company retains the right to have any publication submitted to the Company for review at least 30 days prior to the same paper being submitted for publication or presentation. Investigators must undertake not to submit any part of their individual data for publication without the prior consent of LEO.